CLINICAL TRIAL: NCT02939768
Title: Effects of High-intensity Interval Training and/or Strength Training on Inflammatory, Oxidative Stress and Glycemic Metabolism Parameters in Type 1 Diabetes Mellitus Patients
Brief Title: Impact of Different Types of Exercise Training on Biochemical Markers of Insulin-dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53935916.9.0000.5347
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training protocols (Experimental): Participants will be randomized in one of three groups: HIIT, ST or ST combined with HIIT (ST+HIIT). Each training protocol will last 10 weeks, being the initial two weeks designed to participants' gradual adaptations to respective training protocol, with sessions performed three times per week in non-consecutive days.
  Interventions: Other: High-intensity interval training (HIIT); Other: Strength training (ST); Other: ST combined with HIIT (ST+HIIT)
- Control period (No Intervention): Before interventions (exercise training protocols), all participants will participate of a control period lasting one month, where participants will be encouraged to maintain their habitual lifestyle and usual diet habits.

INTERVENTIONS:
Other: High-intensity interval training (HIIT) — The HIIT sessions will be performed on cycle ergometers and will be consisted of 10 x 60-s cycling intervals interspersed with 60 s recovery. Individual workloads will be selected to elicit ~90% maximal heart rate attained in the cardiorespiratory fitness test (HRmax). A passive or active recovery will be given among high-intensity stimulus. Each training session will include 3-min warm-up and 2-min cool-down phase performed ~50% (HRmax), totalling 25 min. This intervention will last 10 weeks.
  Arms: Exercise training protocols
Other: Strength training (ST) — ST protocol will consist of three sets performed at maximum weight that participants could move eight times with good technique in the following exercises: supine bench press (pectoralis major), leg press (quadriceps, biceps femoris, gluteus maximus), lat pulldown (latissimus dorsi), leg extension (quadriceps), shoulder press (deltoids), leg curl (biceps femoris) and abdominal crunch (abdominal muscles). It will be given 1-min rest between series, totalizing approximately 35 min of ST. This intervention will last 10 weeks.
  Arms: Exercise training protocols
Other: ST combined with HIIT (ST+HIIT) — Participants in the ST+HIIT group will execute ST and HIIT (in this order) above described in the same training session, lasting approximately 60 min. This intervention will last 10 weeks.
  Arms: Exercise training protocols

SUMMARY:
Background: Type 1 diabetes mellitus (T1DM) is characterized by the destruction of β cells and consequent loss of insulin secretion due an autoimmune process, being associated with increased cardiovascular risk, oxidative stress and inflammation.

Considering that most people with T1DM do not reach recommended levels of physical activity due to concern about the rapid drop in blood sugar and the excuse of "lack of time", shorter sessions of exercise that provide several benefits should be encouraged. Thus, this work aims to compare the effects of high-intensity interval training (HIIT), strength training (ST) and both interventions on several blood markers and functional parameters in T1DM patients.

Study hypothesis: (1) ST+HIIT will be more beneficial than HIIT, which in turn will be more beneficial than ST, on modification of blood levels of pro and anti-inflammatory, pro and antioxidant, lipid, renal and glucose metabolism parameters and (2) ST+HIIT will be more beneficial than HIIT, which in turn will be more beneficial than ST, on modification of functional parameters, body composition and maximal oxygen uptake.

DETAILED DESCRIPTION:
Background: Type 1 diabetes mellitus (T1DM), which represents 5-10% of total cases of diabetes mellitus, is characterized by the destruction of β cells and consequent loss of insulin secretion due a autoimmune process. In diabetic patients, micro (nephropathy, neuropathy and retinopathy) and macrovascular (coronary arterial disease, peripheral artery disease, stroke) complications are major causes of morbidity and mortality. It is recommended that diabetics perform at least 150 minutes (min) per week of moderate aerobic exercise divided into at least three days per week, in addition to performing strength training (ST) on two or more days of the week. Considering that most people with T1DM do not reach recommended levels of physical activity due the fear of hypoglycemia and "lack of time", shorter sessions of exercise that provide several benefits should be encouraged. Conversely, reviews studies have demonstrated that sessions composed by ST exercises or high-intensity interval exercise (HIIE) reduce the risk of hypoglycemia during or after the physical effort, when compared with continuous aerobic exercise in T1DM patients, probably via increased hepatic glucose production and transitory inhibition of peripheral glucose uptake. The high-intensity interval training (HIIT) is known by improving glycemic control and muscular adaptations on lipid metabolism in type 2 diabetes mellitus patients, although no studies have used this model of training in T1DM individuals.

Methods: Twenty-seven sedentary T1DM patients (18-40 yo) will be recruited to this randomized clinical trial. Volunteers will sign an informed written consent before enrollment in the study, which was approved by the Ethics Committee of Federal University of Rio Grande do Sul. Initially, all individuals will participate of a control period lasting four weeks, in which they will be asked to maintain their habitual level of physical activity and the usual eating pattern. After, participants will be randomized in three groups: HIIT, ST or ST+HIIT, each lasting ten weeks, with training sessions performed three times/week in cycle ergometers and/or weight machines. HIIT protocol will be consisted of 10 x 1 min cycling bouts performed ~90% maximal heart rate interspersed with 1 min active recovery. ST will consist of three sets performed at the subjects' 10 repetitions maximum load in seven exercises. Participants in the ST+HIIT will perform both training protocols in the same session.

Before control period and before and after interventions, submaximal strength tests, cardiorespiratory fitness test, 3-day diet record and blood draws will be assessed/performed. Body composition will be evaluated before and after the training period. At the 4th week of interventions, the submaximal strength tests and cardiorespiratory fitness test will be assessed for adjusting loads.

According the normality of data, paired Student's t test or Wilcoxon signed rank test will be utilized to determine differences before and after control period. The homogeneity of variances will be confirmed by Mauchly's test, and a Greenhouse-Geisser correction will be applied to the degrees of freedom if the sphericity assumption is violated. Blood outcomes, maximal oxygen uptake and strength values will be analyzed using a two-way ANOVA (3 conditions vs 2 times) with repeated-measures and subsequent Bonferroni post hoc analysis when required. Statistical Package for Social Sciences (SPSS 19.0 Inc, Chicago, USA) will be utilized and statistical significance set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c < 10%;
* Have lived with T1DM for at least four years;
* Physically inactive status (< 150 min of self-reported structured physical activity per week in the previous three months).

Exclusion Criteria:

* Creatinine > 1,3 mg/dL;
* Cardiovascular diseases;
* Retinopathy;
* Severe musculoskeletal injuries;
* Recent infections;
* Use of antioxidant supplements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | End of 10-week exercise period
  HbA1c levels will be determined in the automated analyzer.
Tumor necrosis factor alpha (TNF-α) | End of 10-week exercise period
  The plasma levels of TNF-α will be determined by enzyme-linked immunosorbent assay using commercial kits for human, according to manufacturer's instructions.
Mitochondrial superoxide dismutase (MnSOD) activity | End of 10-week exercise period
  MnSOD isoform activity will be measured spectrophotometrically in mononuclear cells supernatants, according to a method previously described.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- [Derived] Farinha JB, Ramis TR, Vieira AF, Macedo RCO, Rodrigues-Krause J, Boeno FP, Schroeder HT, Muller CH, Boff W, Krause M, De Bittencourt PIH Jr, Reischak-Oliveira A. Glycemic, inflammatory and oxidative stress responses to different high-intensity training protocols in type 1 diabetes: A randomized clinical trial. J Diabetes Complications. 2018 Dec;32(12):1124-1132. doi: 10.1016/j.jdiacomp.2018.09.008. Epub 2018 Sep 19. PMID 30270019